CLINICAL TRIAL: NCT05240664
Title: Effects of An Advance Care Planning Programme for Persons With Early Dementia And Their Family Caregivers in the Community
Brief Title: Effects of An ACP Programme for Older People With Early Dementia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hong Kong Metropolitan University (Other)
Collaborators: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Ms Cheryl Yeung Chi Yan, Principal Investigator, Hong Kong Metropolitan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: CREC 2019.438
Record Dates: First submitted 2022-01-19; First posted 2022-02-15 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Dementia, Mild
Keywords: advance care planning
MeSH Terms: conditions — Dementia; Lymphoma, Follicular

STUDY DESIGN:
Intervention Model Description: Dyads of participants recruited from all elderly community centres will be randomized at block size equals to 4 in 1:1 ratio into intervention group and control group.
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors will be blinded to the group assignment and research question.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACP intervention (Experimental): It is a theory-driven ACP programme specifically designed for PWEDs and their family caregivers. The intervention is underpinned by the Bandura's self-efficacy model.
  Interventions: Behavioral: Have A Say Programme
- Attention-control health talks (Placebo Comparator): Dyads of participants in the control group will receive health talks. This is to differentiate the effect of the intervention from the effect of the extra time and attention given to the participants.
  Interventions: Behavioral: Attention-control health talks

INTERVENTIONS:
Behavioral: Have A Say Programme — Each dyad of participants will receive a 4-session ACP programme, which consists of 2 group-based sessions and 2 dyadic sessions, one hour for each session. The group-based sessions are led by nurse which include didactic educational components, guided reflection, videos, and group sharing. Dyads of participants will be provided with information about ACP, the trajectory of dementia, their future healthcare needs and caring options. Their values and care preferences on future care will be elicited in a consistent manner. The dyadic sessions are facilitated by trained ACP facilitators and guided by an ACP booklet. Dyads of participants will be supported to have an individualized ACP discussion guided by an ACP booklet. By the end of the programme, each dyad of participants will be given an ACP booklet documenting the ACP process.
  Arms: ACP intervention
Behavioral: Attention-control health talks — Dyads of participants in the control group will receive 4-session health talks. One hour for each session, and once weekly. The contents of the health talks are neither dementia-specific nor related to ACP, and cover general health information for elderly, such as drug safety, home safety, exercise and health, and healthy diet.
  Arms: Attention-control health talks

SUMMARY:
Advance care planning (ACP) has been widely advocated for persons with early stage dementia (PWEDs). This proposed study attempts to promote the uptake of ACP for this population and their family caregivers in the community and to examine the effects of an ACP programme "Have a Say" for this population. It is hypothesized that participants in the intervention group will be more engaged in ACP and their dyadic concordance on end-of-life care preference with their family caregivers will be significantly higher than that in the control group.

DETAILED DESCRIPTION:
This study aims to evaluate the effects of an advance care planning (ACP) programme "Have a Say" for persons with early stage dementia (PWEDs) and their family caregivers in the community. A randomized controlled trial with repeated blinded outcome assessment will be conducted to assess the effects of an ACP programme on dyads of PWEDs and their family caregivers recruited from elderly community centres. Individuals who have a clinical diagnosis of any form of dementia at the early stage or have a Global Deterioration Score (GDS) 3 or 4 will be eligible to this study. Participants in the experimental group will receive a 4-session ACP programme. It includes an educational component, guided reflection and ACP discussion through a series of group-based activity and dyadic discussion delivered by trained ACP facilitator and guided by an ACP booklet. Dyads of participants will be provided with information about the trajectory of dementia, their future healthcare needs and caring options. Their values and care preferences on future care will be elicited in a consistent manner. They will be supported to have an individualized ACP discussion. Individuals assigned to the control group will receive attention-control health talks. The primary study outcome is the ACP engagement level of PWEDs. Secondary outcome is the dyadic concordance on end-of-life care preference. Adverse outcomes such as depression and caregivers' burden will also be evaluated. Data collection will be conducted at baseline, immediately after, and one-month after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* being Chinese,
* being a Cantonese speaker,
* having a formal diagnosis of any form of dementia at the early stage, or having a Global Deterioration Scale score 3-4,
* having a designated family caregiver in direct contact and willing to participate in this study.

Exclusion Criteria:

* non-communicable,
* mentally incompetent,
* received an ACP intervention,
* have previously signed an advance directive,
* have other life-limiting chronic illnesses.

A family caregiver involved in primary responsibility for caring and care-related decisions for the PWED will also be recruited. Paid caregivers are to be excluded.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-01-09 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Change in advance care planning engagement | Outcome will be measured at baseline, immediately after intervention, and 1-month after
  The validated 9-item Advance Care Planning (ACP) Engagement Survey will be used to measure the engagement of PWED in the ACP process. Each item is measured on a five-point Likert scale and average 5-point scores will be calculated. It is originated from a longer version of 82 items measuring factors affecting the process of ACP engagement, including knowledge, contemplation, self-efficacy, and readiness. This shorter version reported sound psychometric properties and able to detect change across a broad range of ACP behaviours and ACP domains, with Cronbach's alpha =0.84, cross-sectional correlations =0.85, and delta correlations =0.68. The Chinese version of the ACP Engagement Survey is validated and reported sound psychometrical properties. This scale is composed of self-efficacy subscale and readiness subscale. Higher score reflects a higher level of ACP engagement.

SECONDARY OUTCOMES:
Change in dyadic concordance of preference on end-of-life care | Outcome will be measured at baseline, immediately after intervention, and 1-month after
  The Life-Support Preferences Questionnaire will be used to measure the congruence on end-of-life care preferences between each participant dyad. This questionnaire has been modified and validated in the local context. The modified Chinese version of the Life Support Preferences Questionnaire was simplified to assess preferences regarding (i) three kinds of life-sustaining treatments (cardiopulmonary resuscitation, mechanical ventilator and tube feeding) based on three options (want to attempt, refuse or uncertain) and (ii) care goals (comfort-oriented, prolongation of life at all costs or uncertain) regarding a hypothetical end-of-life scenario (terminally ill). This scenario is based on the local advance directive form. Each member of the participated dyad will complete this questionnaire individually simultaneously. Higher score reflects a higher level of dyadic concordance.
change in depression | Outcome will be measured at baseline, immediately after intervention, and 1-month after
  The Cornell Scale for Depression in Dementia will be used to measure the signs and symptoms of depression of PWEDs. It is a validated instrument for various severity levels of dementia patients. This is a 19-item instrument that uses information from interviews with family caregivers. The Chinese version of this instrument reported an expert content validity index as 0.92, and its concurrent validity with the Geriatric Depression Scale short form is 0.322 (p<0.001). Its Cronbach's alpha for internal consistency reliability is 0.84. Higher score reflects a higher level of depression.
Change in caregivers' stress | Outcome will be measured at baseline, immediately after intervention, and 1-month after
  The Zarit Caregiver Burden Interview (ZBI) will be used to measure the caregivers' stress. It has 12 items. The Cantonese short version of this instrument reported sound psychometric properties. Higher score reflects a higher level of caregivers' stress.

CONTACTS AND LOCATIONS:
Locations (6):
- Hong Kong (6):
  - HKSKH Lok Man Alice Kwok Integrated Service Centre, Kowloon
  - Hong Kong Christian Service, Kowloon
  - Hong Kong Sheng Kung Hui Chuk Yuen Canon Martin District Elderly Community Centre, Kowloon
  - Yang Memorial Methodist Social Service Choi Hung Community Centre for Senior Citizens, Kowloon
  - Jockey Club Centre for Positive Ageing, Shatin
  - Yau On Lutheran Centre for the Elderly, Tuenmen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sudore RL, Heyland DK, Barnes DE, Howard M, Fassbender K, Robinson CA, Boscardin J, You JJ. Measuring Advance Care Planning: Optimizing the Advance Care Planning Engagement Survey. J Pain Symptom Manage. 2017 Apr;53(4):669-681.e8. doi: 10.1016/j.jpainsymman.2016.10.367. Epub 2016 Dec 29. PMID 28042072
- [Background] Sudore RL, Lum HD, You JJ, Hanson LC, Meier DE, Pantilat SZ, Matlock DD, Rietjens JAC, Korfage IJ, Ritchie CS, Kutner JS, Teno JM, Thomas J, McMahan RD, Heyland DK. Defining Advance Care Planning for Adults: A Consensus Definition From a Multidisciplinary Delphi Panel. J Pain Symptom Manage. 2017 May;53(5):821-832.e1. doi: 10.1016/j.jpainsymman.2016.12.331. Epub 2017 Jan 3. PMID 28062339
- [Background] Liu L, Zhao YY, Zhang LH, Chan HY. Measuring Self-Efficacy and Readiness for Advance Care Planning in Chinese Older Adults. J Pain Symptom Manage. 2020 Sep;60(3):622-629. doi: 10.1016/j.jpainsymman.2020.06.013. Epub 2020 Jun 20. PMID 32574659
- [Background] Ditto PH, Danks JH, Smucker WD, Bookwala J, Coppola KM, Dresser R, Fagerlin A, Gready RM, Houts RM, Lockhart LK, Zyzanski S. Advance directives as acts of communication: a randomized controlled trial. Arch Intern Med. 2001 Feb 12;161(3):421-30. doi: 10.1001/archinte.161.3.421. PMID 11176768
- [Background] Chan HY, Ng JS, Chan KS, Ko PS, Leung DY, Chan CW, Chan LN, Lee IF, Lee DT. Effects of a nurse-led post-discharge advance care planning programme for community-dwelling patients nearing the end of life and their family members: A randomised controlled trial. Int J Nurs Stud. 2018 Nov;87:26-33. doi: 10.1016/j.ijnurstu.2018.07.008. Epub 2018 Jul 23. PMID 30048916
- [Background] Alexopoulos GS, Abrams RC, Young RC, Shamoian CA. Cornell Scale for Depression in Dementia. Biol Psychiatry. 1988 Feb 1;23(3):271-84. doi: 10.1016/0006-3223(88)90038-8. PMID 3337862
- [Background] Lin JN, Wang JJ. Psychometric evaluation of the Chinese version of the Cornell Scale for Depression in Dementia. J Nurs Res. 2008 Sep;16(3):202-10. doi: 10.1097/01.jnr.0000387307.34741.39. PMID 18792890
- [Background] Zarit SH, Reever KE, Bach-Peterson J. Relatives of the impaired elderly: correlates of feelings of burden. Gerontologist. 1980 Dec;20(6):649-55. doi: 10.1093/geront/20.6.649. No abstract available. PMID 7203086
- [Background] Tang JY, Ho AH, Luo H, Wong GH, Lau BH, Lum TY, Cheung KS. Validating a Cantonese short version of the Zarit Burden Interview (CZBI-Short) for dementia caregivers. Aging Ment Health. 2016 Sep;20(9):996-1001. doi: 10.1080/13607863.2015.1047323. Epub 2015 May 27. PMID 26016419